CLINICAL TRIAL: NCT02611193
Title: Efficacy of Manipulative Treatment for Carpal Tunnel Syndrome: a Randomized Clinical Trial
Brief Title: Efficacy of Manipulative Treatment for Carpal Tunnel Syndrome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fundación para el Fomento de la Investigación Sanitaria y Biomédica de la Comunitat Valenciana (Other)
Responsible Party: Principal Investigator, Julio Domenech, MD-PhD, Fundación para el Fomento de la Investigación Sanitaria y Biomédica de la Comunitat Valenciana
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MOM-STC
Record Dates: First submitted 2015-07-23; First posted 2015-11-20 (Estimated); Last update posted 2015-11-20 (Estimated); Status verified 2015-11

CONDITIONS: Carpal Tunnel Syndrome
MeSH Terms: conditions — Carpal Tunnel Syndrome | interventions — Manipulation, Osteopathic

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Manipulative treatment (Experimental): Manipulative Treatment
  Interventions: Procedure: Manipulative treatment
- Simulated manipulative treatment (Sham Comparator): Simulated manipulative treatment
  Interventions: Procedure: Simulated manipulative treatment

INTERVENTIONS:
Procedure: Manipulative treatment — Manipulative treatment as described by the GBMOIM (Grupo Barcelona de Medicina Ortopédica y Manual) will be perform with extension of the transverse carpal ligament maneuver and fascia release maneuver
  Arms: Manipulative treatment
Procedure: Simulated manipulative treatment — Simulated Manipulative Treatment
  Arms: Simulated manipulative treatment

SUMMARY:
Hypothesis: Manipulative treatment can relieve patients of discomfort and dysfunction and then be utilized as a cheap conservative management of CTS. Study design: Two-groups randomized single-blind interventional study.

DETAILED DESCRIPTION:
Background: Carpal Tunnel Syndrome (CTS) is the most common compressive neuropathy in the upper limb. It considerably impairs patient's quality of life and generates important social consequences due to the lost of productivity and the cost of treatments. Both surgical and conservative treatment are utilized for CTS management. Manipulative treatment is a conservative, non-drug and cheap management option which can be proposed, but by now, treatment guidelines and reviews do not recommend it due to lack of evidence to assess his efficacy.

Hypothesis: Manipulative treatment can relieve patients of discomfort and dysfunction and then be utilized as a cheap conservative management of CTS.

Study design: Two-groups randomized single-blind interventional study. Methods: Sixty-six patients reporting CTS symptoms that are confirmed by clinical exam and nerve conduction studies will be included. Participants will be randomized in two arms, one receiving manipulative treatment and one receiving simulated manipulative treatment (1/week for 4 weeks). The main outcome measures will be the DASH questionnaire, the Boston Carpal Tunnel Syndrome Questionnaire, patient estimate on Visual Analog Scale for pain and the EuroQol-5D scale. All outcomes measures will be administrated to participants before the first manipulation, after the last session (4 weeks) and 12 weeks after the baseline measure.

ELIGIBILITY:
Inclusion Criteria:

* Symptoms of canal tunnel syndrome (CTS) : pain, numbness, paresthesia, diminished grip strength
* Electromyography confirming CTS

Exclusion Criteria:

* Previous surgical procedure for CTS in the same wrist
* Possible secondary CTS : hypothyroidism, diabetes mellitus, pregnancy, rheumatologic diseases, neck or shoulder complaints,
* Hand and wrist pathological conditions as previous disease, intervention, traumatism, anatomic abnormalities in shape or size.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2016-05; Primary Completion 2017-01 (Estimated); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
Change in Boston Carpal Tunnel Questionnaire | Baseline, 4 weeks, 12 weeks
  self-administered questionnaire for the assessment of severity of symptoms and functional status in patients who have carpal tunnel syndrome. It has two distinct scales : a symptom-severity scale (11
  - Page 2 of 3 [DRAFT] - items) and a functional-status scale (8 items). It has been validated and demonstrated to show good responsiveness and reliability in evaluating outcome after carpal tunnel release. The Spanish version has been validated

SECONDARY OUTCOMES:
Change in DASH Outcome Measure | Baseline, 4 weeks, 12 weeks
  30-item, self-report questionnaire designed to measure physical function and symptoms in people with a musculoskeletal disorder of the upper limb. It showed a large degree of responsiveness after CTS treatment and the Spanish version has been validated
Change in Visual Analog Scale for pain | Baseline, 4 weeks, 12 weeks
  VAS has eleven points from 0 to 10, being 0 no pain at all, and 10 the worst pain could ever be imagined
Change in EuroQol-5D scale | Baseline, 4 weeks, 12 weeks
  Quality-of-life's measure instrument which consists of a combination of a 5 items questionnaire and a Visual analogue scale. Both validity and responsiveness have been demonstrated in patients with chronic pain, and it has been evaluated in patients with CTS symptoms. The Spanish version has been validated
Change in strength (Dynamometer) | Baseline, 4 weeks, 12 weeks
  Measuring pulp pinch strength with digits I and II

CONTACTS AND LOCATIONS:
Overall Officials: Julia Schmitt, PM&RResident, Principal Investigator — Hospital Arnau de Vilanova, Valencia, Spain; Julio Domenech, MD-PhD, Study Director — Hospital Arnau de Vilanova, Valencia, Spain